CLINICAL TRIAL: NCT04036292
Title: Multicenter, Randomized, Controlled, Double-Masked, Clinical Trial to Evaluate the Efficacy and Safety of OC-01 (Varenicline) Nasal Spray on Signs and Symptoms of Dry Eye Disease (The ONSET-2 Study)
Brief Title: Evaluation of the Efficacy and Safety of OC-01 Nasal Spray on Signs and Symptoms of Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPP-101
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-08

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Varenicline; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OC-01 Low Dose, 0.6 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, 0.6 mg/ML
  Interventions: Drug: OC-01 (varenicline) nasal spray
- OC-01 High Dose, 1.2 mg/mL (Active Comparator): OC-01 (varenicline) nasal spray, 1.2 mg/ML
  Interventions: Drug: OC-01 (varenicline) nasal spray
- Placebo (vehicle) nasal spray (Placebo Comparator): Placebo (vehicle) nasal spray
  Interventions: Drug: Placebo (vehicle) nasal spray

INTERVENTIONS:
Drug: OC-01 (varenicline) nasal spray — OC-01 (varenicline) nasal spray
  Arms: OC-01 High Dose, 1.2 mg/mL; OC-01 Low Dose, 0.6 mg/mL
Drug: Placebo (vehicle) nasal spray — Placebo (vehicle) nasal spray
  Arms: Placebo (vehicle) nasal spray

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of OC-01 Nasal Spray as compared to placebo on signs and symptoms of dry eye disease.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, controlled, double-masked (including subjects, Investigators, study site personnel, and Sponsor personnel) study designed to evaluate the safety and efficacy of OC-01 (varenicline) nasal spray 0.6 mg/mL and 1.2 mg/mL in adult participants with DED. The study randomized 758 subjects at least 22 years of age with a physicians' diagnosis of DED and meeting all other study eligibility criteria to receive OC-01 (varenicline) nasal spray or placebo twice daily (BID) for 28 days with three additional long-term follow-up visits at 6 weeks, 6 months, and 12 months. Participants who terminated from the study during the treatment period were asked to complete safety assessments (if the participants agree) prior to study exit. Participants who were terminated early from the study were not replaced

ELIGIBILITY:
Inclusion Criteria:

- Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to Visit 1

Exclusion Criteria:

* Have had any intraocular surgery (such as cataract surgery) or extraocular surgery in either eye within three months or refractive surgery (e.g. laser-assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy or corneal implant) within twelve months of Visit 1.
* Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment and mild meibomian gland disease that are typically associated with dry eye disease are allowed.
* Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
* Have a known hypersensitivity to any of the procedural agents or study drug components
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Phoenix, Phoenix, Arizona
  - New Port Beach, Newport Beach, California
  - Fort Collins, Fort Collins, Colorado
  - Waterbury, Waterbury, Connecticut
  - Delray Beach, Delray Beach, Florida
  - Indianapolis, Indianapolis, Indiana
  - Louisville, Louisville, Kentucky
  - Raynham, Raynham, Massachusetts
  - Las Vegas, Las Vegas, Nevada
  - Raleigh, Raleigh, North Carolina
  - Shelby, Shelby, North Carolina
  - Fargo, Fargo, North Dakota
  - Cranberry Township, Cranberry Township, Pennsylvania
  - Warwick, Warwick, Rhode Island
  - Sioux Falls, Sioux Falls, South Dakota
  - Nashville, Nashville, Tennessee
  - Austin, Austin, Texas
  - Houston, Houston, Texas
  - San Antonio, San Antonio, Texas
  - Layton, Layton, Utah
  - Lynchburg, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hauswirth SG, Kabat AG, Hemphill M, Somaiya K, Hendrix LH, Gibson AA. Safety, adherence and discontinuation in varenicline solution nasal spray clinical trials for dry eye disease. J Comp Eff Res. 2023 Jun;12(6):e220215. doi: 10.57264/cer-2022-0215. Epub 2023 Apr 25. PMID 37096956
- [Derived] Nijm LM, Zhu D, Hemphill M, Blemker GL, Hendrix LH, Kabat AG, Gibson AA. Does Menopausal Status Affect Dry Eye Disease Treatment Outcomes with OC-01 (Varenicline Solution) Nasal Spray? A Post Hoc Analysis of ONSET-1 and ONSET-2 Clinical Trials. Ophthalmol Ther. 2023 Feb;12(1):355-364. doi: 10.1007/s40123-022-00607-7. Epub 2022 Nov 18. PMID 36401081
- [Derived] Wirta D, Vollmer P, Paauw J, Chiu KH, Henry E, Striffler K, Nau J; ONSET-2 Study Group. Efficacy and Safety of OC-01 (Varenicline Solution) Nasal Spray on Signs and Symptoms of Dry Eye Disease: The ONSET-2 Phase 3 Randomized Trial. Ophthalmology. 2022 Apr;129(4):379-387. doi: 10.1016/j.ophtha.2021.11.004. Epub 2021 Nov 10. PMID 34767866

RESULTS

PARTICIPANT FLOW:
Groups:
- OC-01 Low Dose 0.6 mg/mL BID for 28 Days: OC-01 (varenicline) nasal spray, 0.6 mg/ML BID for 28 days
- OC-01 High Dose 1.2 mg/mL BID for 28 Days: OC-01 (varenicline) nasal spray 1.2 mg/mL BID for 28 days
- Placebo BID for 28 Days: Placebo (vehicle) nasal spray BID for 28 days
Period: Overall Study
Arm/Group | OC-01 Low Dose 0.6 mg/mL BID for 28 Days | OC-01 High Dose 1.2 mg/mL BID for 28 Days | Placebo BID for 28 Days
Started | 260 | 246 | 252
Completed | 239 | 212 | 228
Not Completed | 21 | 34 | 24

BASELINE CHARACTERISTICS:
Population: Subjects in the ITT population
Groups:
- OC-01 Low Dose 0.6 mg/mL BID for 28 Days: OC-01 (varenicline) nasal spray, 0.6 mg/ML BID for 28 days
  OC-01 (varenicline) nasal spray: OC-01 (varenicline) nasal spray
- OC-01 High Dose 1.2 mg/mL BID for 28 Days: OC-01 (varenicline) nasal spray, 1.2 mg/ML BID for 28 days
  OC-01 (varenicline) nasal spray: OC-01 (varenicline) nasal spray
- Placebo (Vehicle) Nasal Spray BID for 28 Days: Placebo (vehicle) nasal spray BID for 28 days
  Placebo (vehicle) nasal spray: Placebo (vehicle) nasal spray
- Total: Total of all reporting groups
Arm/Group | OC-01 Low Dose 0.6 mg/mL BID for 28 Days | OC-01 High Dose 1.2 mg/mL BID for 28 Days | Placebo (Vehicle) Nasal Spray BID for 28 Days | Total
Number analyzed (Participants) | 260 | 246 | 252 | 758
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (12.76) | 58.4 (13.03) | 58.4 (13.29) | 58.8 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 181 | 201 | 576
  Male | 66 | 65 | 51 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 37 | 36 | 100
  Not Hispanic or Latino | 233 | 209 | 216 | 658
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 2 | 6 | 9
  Race: Asian | 11 | 7 | 5 | 23
  Race: Black or African American | 27 | 35 | 29 | 91
  Race: Native Hawaiian or other Pacific Islander | 2 | 0 | 1 | 3
  Race: White | 219 | 200 | 211 | 630
  Race: Other | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 260 | 246 | 252 | 758
Baseline Schirmer's Test Score (mm) [Mean (Standard Deviation); unit: mm] — Schirmer's test score from 0-35 mm where a higher score is indicative of a better outcome.
  mm | 5.1 (2.95) | 5.4 (2.93) | 4.9 (2.89) | 5.1 (2.93)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Achieve ≥10 mm Improvement in Schirmer's Test Score From Baseline at Visit 4 (Day 28)
Description: The primary endpoint was the percentage of subjects who achieve ≥10 mm improvement in Schirmer's Test Score from baseline to 28 days in the study eye following treatment with OC-01. Schirmer's test scores from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: 28 Days [Visit 1 (baseline) and Visit 4b (28 days)]
Population: Subjects in the ITT-LOCF population
Measure: Count of Participants; unit: Participants
Groups:
- OC-01 Low Dose, 0.6 mg/mL: OC-01 (varenicline) nasal spray, 0.6 mg/ML
  OC-01 (varenicline) nasal spray
- OC-01 High Dose, 1.2 mg/mL: OC-01 (varenicline) nasal spray, 1.2 mg/ML
  OC-01 (varenicline) nasal spray
Arm/Group | OC-01 Low Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo (Vehicle) Nasal Spray
Number analyzed (Participants) | 260 | 246 | 252
Participants | 123 | 121 | 70

2. Secondary Outcome: Mean Change From Baseline in Eye Dryness Score in CAE at Week 4 at 5 Minutes
Description: Change in Eye Dryness Score Eye from baseline in CAE at 4 Weeks at 5 minutes post treatment. Eye dryness score on a Visual Analogue Scale (VAS) from 0 (no dryness) to 100 (maximum dryness) millimeters where a lower score is indicative of a better outcome.
Time Frame: 28 Days [Visit 1 (baseline) and Visit 4a (28 days)]
Population: Subjects in the mITT-2 population
Measure: Least Squares Mean (Standard Error); unit: mm
Groups:
- Placebo: Placebo (vehicle) nasal spray
Arm/Group | OC-01 Low Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 187 | 171 | 169
mm | -10.3 (1.62) | -9.0 (1.75) | -7.4 (1.74)

3. Secondary Outcome: Mean Change From Baseline in Eye Dryness Score From Baseline to Day 28
Description: Change in Eye Dryness Score Eye from baseline to 28 days. Eye dryness score on a Visual Analogue Scale (VAS) from 0 (no dryness) to 100 (maximum dryness) millimeters where a lower score is indicative of a better outcome.
Time Frame: 28 Days [Visit 1 (baseline) and Visit 4b (28 days)]
Population: Subjects in the ITT-LOCF population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | OC-01 Low Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 255 | 242 | 248
mm | -19.8 (1.54) | -22.2 (1.61) | -15.4 (1.57)

4. Secondary Outcome: Mean Change Form Baseline in Schirmer's Test Score From Baseline to Day 28
Description: Change in Schirmer test score from baseline to Day 28. Schirmer's test scores from 0-35 mm where a higher score is indicative of a better outcome.
Time Frame: 28 Days [Visit 1 (baseline) and Visit 4b (28 days)]
Population: Subjects in the ITT-LOCF population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | OC-01 Low Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 251 | 235 | 248
mm | 11.3 (0.61) | 11.5 (0.64) | 6.3 (0.61)

5. Secondary Outcome: Mean Change From Baseline in Eye Dryness Score in the Study Eye at Week 2
Description: Chang in Eye Dryness Score Eye from baseline to 28 days. Eye dryness score on a Visual Analogue Scale (VAS) from 0 (no dryness) to 100 (maximum dryness) millimeters where a lower score is indicative of a better otucome.
Time Frame: 14 Days [Visit 1 (baseline) and Visit 3 (14 days)]
Population: Subjects in the ITT-LOCF population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | OC-01 Low Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 255 | 239 | 248
mm | -16.5 (1.38) | -17.9 (1.45) | -12.7 (1.41)

6. Secondary Outcome: Mean Change From Baseline in Eye Dryness Score in the Study Eye at Week 1
Description: as for outcome 3
Time Frame: 7 Days [Visit 1 (baseline) and Visit 2 (7 days)]
Population: Subjects in the ITT population
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | OC-01 Low Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo
Number analyzed (Participants) | 254 | 239 | 248
mm | -15.7 (1.33) | -15.4 (1.40) | -13.3 (1.35)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug administration until the final study visit at Visit 7
Arm/Group | OC-01 Low Dose, 0.6 mg/mL | OC-01 High Dose, 1.2 mg/mL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/260 | 2/245 | 1/251
Serious Adverse Events (participants affected / at risk) | 5/260 | 12/245 | 9/251
Other Adverse Events (participants affected / at risk) | 253/260 | 243/245 | 158/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC-01 Low Dose, 0.6 mg/mL (N=260) | OC-01 High Dose, 1.2 mg/mL (N=245) | Placebo (N=251)
Coronavirus infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0 | 1
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 1
Hip surgery (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC-01 Low Dose, 0.6 mg/mL (N=260) | OC-01 High Dose, 1.2 mg/mL (N=245) | Placebo (N=251)
conjunctival hyperaemia (Eye disorders) | 12 | 11 | 7
Visual acuity reduced (Eye disorders) | 9 | 9 | 11
Blepharitis (Eye disorders) | 3 | 1 | 3
Pinguecula (Eye disorders) | 1 | 3 | 2
Cataract (Eye disorders) | 2 | 0 | 3
Conjunctival haemorrage (Eye disorders) | 1 | 1 | 3
Eye irritation (Eye disorders) | 1 | 1 | 3
Posterior capsule opacification (Eye disorders) | 0 | 2 | 3
Meibomian gland dysfunction (Eye disorders) | 1 | 2 | 1
Cataract nuclear (Eye disorders) | 1 | 1 | 1
Eye pruritus (Eye disorders) | 1 | 2 | 0
Lacrimation increased (Eye disorders) | 1 | 1 | 1
Arcus lipoides (Eye disorders) | 0 | 1 | 1
Chalazion (Eye disorders) | 1 | 0 | 1
Conjunctival disorder (Eye disorders) | 1 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 1
Erythema of eyelid (Eye disorders) | 1 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 1
Ocular hyperaemia (Eye disorders) | 0 | 2 | 0
Punctate keratitis (Eye disorders) | 1 | 0 | 1
Swelling of eyelid (Eye disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1
Cataract subcapsular (Eye disorders) | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 1 | 0
corneal epithelium defect (Eye disorders) | 0 | 1 | 0
corneal opacity (Eye disorders) | 1 | 0 | 0
Diabetic retinal oedema (Eye disorders) | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 1 | 0
Ectropion (Eye disorders) | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0
Eyelid cyst (Eye disorders) | 1 | 0 | 0
Eyelid margin crusting (Eye disorders) | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Glare (Eye disorders) | 1 | 0 | 0
Keratopathy (Eye disorders) | 0 | 0 | 1
Macular hole (Eye disorders) | 1 | 0 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Trichiasis (Eye disorders) | 1 | 0 | 0
Visual impairement (Eye disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 3 | 2 | 2
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0 | 0
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Melanocytic maevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 247 | 237 | 73
Cough (Respiratory, thoracic and mediastinal disorders) | 49 | 54 | 5
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 35 | 44 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 12
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 9
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 2
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 9 | 16 | 14
Sinusitis (Infections and infestations) | 0 | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 0
Influenza (Infections and infestations) | 1 | 3 | 3
Urinary tract infection (Infections and infestations) | 2 | 1 | 3
Bronchitis (Infections and infestations) | 3 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 3
Instillation site irritation (General disorders) | 21 | 36 | 3
Headache (Nervous system disorders) | 8 | 7 | 3
Dysgeusia (Nervous system disorders) | 4 | 5 | 0
Migraine (Nervous system disorders) | 3 | 1 | 2
Dizziness (Nervous system disorders) | 3 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Coronavirus test positive (Investigations) | 3 | 4 | 2
Hypertension (Vascular disorders) | 4 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT04036292/Prot_002.pdf
  • Statistical Analysis Plan (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT04036292/SAP_003.pdf